CLINICAL TRIAL: NCT04406376
Title: Do We Need to Taper Down Steroid Therapy for Bell's Palsy: A Prospective Randomized Controlled Trial
Brief Title: Do We Need to Taper Down Steroid Therapy for Bell's Palsy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Carmel Medical Center (Other)
Responsible Party: Principal Investigator, Itai Margulis, Intern, Department of Otolaryngology Head and Neck Surgery, Principal Investigator, Medical Doctor, Carmel Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMC-20-0001-CTIL
Record Dates: First submitted 2020-05-09; First posted 2020-05-28 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Bell Palsy
Keywords: Tapering Down; Adverse Effects; House Brackmann; Steroids; Prednisone
MeSH Terms: conditions — Bell Palsy | interventions — Prednisone

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to recieve one of the following steroids regimens:
  1. Prednisone 1 mg/kg (max. 60 mg) daily for 7 days, 40 mg for 2 days, 20 mg for 2 days (Total 11 days)
  2. Prednisone 1 mg/kg (max. 60 mg) daily for 7 days (Total 7 days)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tapering Down of Steroids (Active Comparator): Prednisone 1 mg/kg (max. 60 mg) daily for 7 days, 40 mg for 2 days, 20 mg for 2 days (Total 11 days)
  Interventions: Drug: Prednisone tablet
- No Tapering Down of Steroids (Active Comparator): Prednisone 1 mg/kg (max. 60 mg) daily for 7 days (Total 7 days)
  Interventions: Drug: Prednisone tablet

INTERVENTIONS:
Drug: Prednisone tablet — Treatment of Bell's Palsy with prednisone, with or without tapering down.

SUMMARY:
Bell's palsy [BP] is defined as acute idiopathic peripheral facial palsy or paralysis.

Additional symptoms frequently include pain around or behind the ear, impaired tolerance to ordinary levels of noise and disturbed sense of taste on the same side. It affects men and women more or less equally.

There is a consensus in the literature regarding the importance of steroid treatment for improving recovery rates and sequela of BP. Moreover, there is increasing level of high quality of evidence in recent years for a combined antiviral and steroids treatment for severe BP (House Brackmann [HB] 5-6).

Adverse effects (AEs) were reported in 1-12% of patients treated with steroids, antivirals or placebo. The AEs reported were dyspepsia, loss of blood sugar control, headache, fatigue, dizziness and insomnia, recurrent duodenal ulcers, mood swings, and acute psychosis. All effects resolved when treatment was stopped.

Although steroid and antivirals are widely used for BP, there is a high variability of steroids treatment, both in the dosage given and in the way of tapering down.

Among the different steroid regimens used were: prednisone 1 mg/kg for 5 days tapered to 10 mg/day for remaining 5 days; prednisone (1 mg/kg for 10 days then tapered to zero over the next 6 days); prednisolone 60 mg for 5 days, 30 mg for 3 days, and 10 mg for 2 days.

House-Brackmann (HB) system is widely used for facial function assessment. It is based on a six-grade score, where grade I is normal function, grade VI is complete absence of facial motor function, and grades II to V are intermediate.

Steroid-induced side effects generally require tapering of the drug as soon as the disease being treated is under control. Tapering must be done carefully to avoid both recurrent activity of the underlying disease and possible cortisol deficiency resulting from hypothalamic-pituitary-adrenal axis (HPA) suppression. However, according to a review by Furst et al (2019), a patient who has received any dose of glucocorticoid for less than 3 weeks or patients treated with alternate-day prednisone at a dose of less than 10 mg (or its equivalent) are unlikely for HPA suppression. They concluded that short-term glucocorticoid therapy (up to three weeks), even if at a fairly high dose, can simply be stopped and need not to be tapered..

According to the above, the investigators assume that a rapid withdrawal of steroids after short course of treatment for BP should neither influence the efficacy or safety of treatment.

Finally, steroid regimen may be hard to follow for some patients and can results in confusion and frustration. Simplifying steroid regimen, such as skipping withdrawal if not necessary, may solve this problem.

The objective of our study is to determine the effectiveness and safety of prednisone treatment with no tapering down for Bell's Palsy.

DETAILED DESCRIPTION:
A prospective randomized controlled trial of adult patients diagnosed with BP in the otolaryngology emergency department within 72 hours of symptoms onset.

Patients will be randomized to receive one of the following steroids regimens:

1. Prednisone 1 mg/kg (max. 60 mg) daily for 7 days, 40 mg for 2 days, 20 mg for 2 days (Total 11 days)
2. Prednisone 1 mg/kg (max. 60 mg) daily for 7 days (Total 7 days)

In addition, both groups will receive the following treatment when indicated:

* Mosturizing eye drops for 14 days or until complete recovery (HB-1)
* Mosturizing eye gel for 14 days or until complete recovery (HB-1)
* Omepradex once daily during prednisone treatment (unless the patient receives chronic treatment with any proton pump inhibitor).
* Acyclovir for 7 days in cases of severe BP (HB 5-6).

Patients' follow-up visits: 14 days, 1 month, 3 months. If recovery will be completed before 1 month, no more follow up visits will be taken.

In addition, side effects of prednisone use will be assessed as well as compliance to therapy and duration of additional symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (≥18 years) diagnosed with BP within 72 hour of onset.
2. Adult patients willing to get treatment, attending follow up visits and signing informed consent.

Exclusion Criteria:

1. Patients treated with antivirals (i.e acyclovir) for any reason simultaneously, such as Herpes Zoster (Ramsay- Hunt syndrome).
2. Palsy onset > 72 hours before diagnosis or unknown onset.
3. Previous episodes of BP.
4. Patients suspected for hypothalamic-pituitary-adrenal (HPA) axis suppression who have to be cautiously tapered due to high risk for adrenal insufficiency: steroid treatment in any dosage for more the 3 weeks (due to other indication) or cushingoid appearance.
5. Contraindication for steroid use: uncontrolled diabetes or hypertension, psychosis, peptic ulcer or upper GI bleeding, liver cirrhosis or portal hypertension, known allergy to prednisone, etc. Any case in which steroid treatment was stopped earlier than planned by the patient or the physician.
6. Any conditions suspicious for non-idiopathic facial palsy: chronic otitis media, acute otitis media, mastoiditis, temporal bone/middle ear trauma, other cranial nerve neuropathies (i.e cranial nerve VIII), cerebrovascular disorders, tumor affecting facial nerve (i.e, parotid malignancy, schwannoma) or systemic causes (i.e multiple sclerosis, meningitis, sarcoidosis, HIV infection, etc).
7. Patients with low compliance for treatment according to the physician.
8. Pregnancy or breast-feeding patients.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2020-05-12 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
House-Brackmann scale | 14 days- 90 days
  Time to complete recovery (Grade I- normal function) of facial palsy using the House-Brackmann scale for assessment. The scale is assessed by an ENT physician in four standard poses: at rest, with a forced smile, with raised eyebrows, and with eyes tightly closed and scored between I (normal function)- VI (complete palsy, worse outcome).

SECONDARY OUTCOMES:
Time to incomplete recovery | 14 days- 90 days
  Time to presentation of House-Brackmann Grade II or worse and the difference between House-Brackmann scores between visits (i.e improvement from House-Brackmann 4 to 2)
Occurrence of Motor Synkinesis | 14 days- 90 days
  Occurrence of abnormal synchronization of facial movement where muscles, other than those intended, contract together during a particular movement pattern.
Duration of neurological symptoms | 14 days- 90 days
  Duration of hypoesthesia (trigeminal/ glossopharyngeal), periauricular pain, dysgusia, hyperacusis
Duration of ocular symptoms | 14 days- 90 days
  Duration of dryness, epiphora, itching, eye pain, etc
Adverse effects of prednisone use | 14 days- 90 days
  Incidence of dyspepsia, loss of blood sugar control, headache, fatigue, dizziness and insomnia, recurrent duodenal ulcers, mood swings, acute psychosis, etc

CONTACTS AND LOCATIONS:
Overall Officials: Yoav Yanir, MD, Study Director — Carmel Medical Center
Locations (1):
- Lady Davies Carmel Medical Center. Department of Otolaryngology, Head and Neck Surgery, Haifa, North, Israel